CLINICAL TRIAL: NCT05765279
Title: An Investigator Initiated Clinical Study To Evaluate the Efficacy and Safety of HH-120 Nasal Spray as Post Exposure Prophylaxis (PEP) Regimen in Adult Close Contacts of Individuals Infected With SARS-CoV-2
Brief Title: A Study to Assess the Efficacy of HH-120 Nasal Spray for Prevention of SARS-CoV-2 Infection in Adult Close Contacts of Individuals Infected With SARS-CoV-2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Beijing Ditan Hospital (Other)
Responsible Party: Principal Investigator, Ronghua Jin, Professor, Beijing Ditan Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: HH120-NS02
Record Dates: First submitted 2023-03-01; First posted 2023-03-13 (Actual); Last update posted 2023-03-13 (Actual); Status verified 2023-03

CONDITIONS: SARS-CoV-2 Infection
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Treatment Group 1 (Experimental)
  Interventions: Drug: HH-120 nasal spray 1
- Treatment Group 2 (Experimental)
  Interventions: Drug: HH-120 nasal spray 2
- Control Group 3 (Placebo Comparator)
  Interventions: Drug: Placebo Comparator 1
- Control Group 4 (Placebo Comparator)
  Interventions: Drug: Placebo Comparator 2

INTERVENTIONS:
Drug: HH-120 nasal spray 1 — HH-120 nasal spray 5 times daily for 3 consecutive days
  Arms: Treatment Group 1
Drug: HH-120 nasal spray 2 — HH-120 nasal spray 8 times daily for 3 consecutive days
  Arms: Treatment Group 2
Drug: Placebo Comparator 1 — Placebo nasal spray 5 times daily for 3 consecutive days
  Arms: Control Group 3
Drug: Placebo Comparator 2 — Placebo nasal spray 8 times daily for 3 consecutive days
  Arms: Control Group 4

SUMMARY:
An Investigator-initiated, Randomized, Single-Blind, Placebo-Controlled Trial to Evaluate the Efficacy of SARS-Cov-2 Post Exposure Prophylaxis and Safety of HH-120 nasal spray

ELIGIBILITY:
Inclusion Criteria:

* Participants aged 18 to 65 years.
* Participants who have close contact with a SARS-CoV-2 infected individual (index case) are required to be randomized within 72 hours upon close contact.
* Willing and able to provide written informed consent, or with a legal representative who can provide informed consent.

Exclusion Criteria:

* Have a history of severe allergy or hyper-sensitivity to inhaled allergen.
* Pregnant or breastfeeding women.
* Have participated, within the last 180 days prior to the screening, in a clinical study involving an investigational intervention of SARS-CoV-2 neutralizing antibody.
* Have other conditions not suitable for the study per investigator's discretion.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 281 (Actual)
Dates: Start 2022-10-20 (Actual); Primary Completion 2022-12-06 (Actual); Study Completion 2022-12-06 (Actual)

PRIMARY OUTCOMES:
Proportion of subjects who have a RT-qPCR confirmed SARS-CoV-2 infection. | Day 1 to Day 10

SECONDARY OUTCOMES:
Proportion of subjects who have a symptomatic RT-qPCR confirmed SARS-CoV-2 infection. | Day 1 to Day 10
Proportion of subjects who have an asymptomatic RT-qPCR confirmed SARS-CoV-2 infection. | Day 1 to Day 10

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Ditan Hospital,Capital Medical University, Beijing, Beijing Municipality, China